CLINICAL TRIAL: NCT02644369
Title: Investigator-initiated Phase II Study of Pembrolizumab Immunological Response Evaluation
Brief Title: Study of the Effects of Pembrolizumab in Patients With Advanced Solid Tumors
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSPIRE-001
Record Dates: First submitted 2015-10-27; First posted 2015-12-31 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Cancer of Head and Neck; Triple Negative Breast Cancer; Epithelial Ovarian Cancer; Malignant Melanoma; Advanced Solid Tumors
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Ovarian Epithelial; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab will be given by intravenous infusion (IV, given by vein) at a dose of 200 mg, once every 3 weeks.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda(TM); MK-3475

SUMMARY:
This is a phase 2 study whose main purpose is to evaluate gene changes and immune biomarkers in patients with solid tumors during treatment with pembrolizumab and in relation to response to treatment.

Pembrolizumab is a monoclonal antibody that is designed to block a protein called programmed cell death 1 ligand 1 (PD-L1) which will allow the body's immune system to kill the cancer cells.

DETAILED DESCRIPTION:
This study will involve treatment with pembrolizumab, tests and procedures done for safety, and the collection of archival tumor tissue, fresh tumor biopsies, and blood samples for biomarker research (including genetic testing).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age or older on day of signing informed consent.
* Have histologically or cytologically-documented, locally-advanced, or metastatic solid malignancy that is incurable and has either (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the patient and treating physician. There is no limit to the number of prior treatment regimens.
* Have one of the following advanced (unresectable and/or metastatic) solid tumor indications:

  * Squamous cell cancer of head and neck
  * Triple negative breast cancer
  * Epithelial ovarian cancer
  * Malignant melanoma
  * Advanced solid tumors
* Have measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Patients for whom newly-obtained samples cannot be provided (e.g. inaccessible or patient safety concern) will not be eligible for this study.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function.
* Negative pregnancy test for female patients of childbearing potential.
* Must use approved methods of birth control during the course of the study and for 120 days after the last dose of study drug.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Study Day 1 or who has not recovered from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in genomic and immune biomarkers that will be measured in blood and tumor pre-treatment, on-treatment and at progression (progression biopsies only done for those who have complete or partial responses, or stable disease for more than 4 months) | 5 years
  T-test or Wilcoxon's test

SECONDARY OUTCOMES:
Overall response rate | 5 years
  summary statistics
Changes in circulating tumor DNA genomic biomarkers | 5 years
  T-test or Wilcoxon's test
Changes in radiomic imaging parameters | 5 years
  T-test or Wilcoxon's test
Correlation between tumor genomic profiles and radiomic imaging signatures | 5 years
  Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Non-parametric tests such as Spearman correlation coefficients, Fisher's exact tests and Wilcoxon rank sum tests may be substituted if necessary.
Changes in immune cell subsets in the blood and tumor microenvironment | 5 years
  T-test or Wilcoxon's test
Positive predictive value and negative predictive value of in vitro predictive assay for Pembrolizumab response | 5 years
  Positive predictive value and negative predictive value
Distribution of drug tumor penetration using a mass spectrometry assay | 5 years
  summary statistics
Baseline tumor RNA expression profile for immune inhibitory genes | 5 years
  summary statistics
Comparison of baseline tumor RNA expression profile for immune inhibitory genes with clinical outcome (response) | 5 years
  T-test or Wilcoxon's test

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hernando-Calvo A, Yang SYC, Vila-Casadesus M, Han M, Liu ZA, Berman AHK, Spreafico A, Razak AA, Lheureux S, Hansen AR, Lo Giacco D, Abbas-Aghababazadeh F, Matito J, Haibe-Kains B, Pugh TJ, Bratman SV, Aleshin A, Berche R, Saavedra O, Garralda E, Elston S, Siu LL, Ohashi PS, Vivancos A, Bedard PL. Combined Transcriptome and Circulating Tumor DNA Longitudinal Biomarker Analysis Associates With Clinical Outcomes in Advanced Solid Tumors Treated With Pembrolizumab. JCO Precis Oncol. 2024 Aug;8:e2400100. doi: 10.1200/PO.24.00100. PMID 39178369
- [Derived] Koppensteiner L, Mathieson L, Pattle S, Dorward DA, O'Connor R, Akram AR. Location of CD39+ T cell subpopulations within tumors predict differential outcomes in non-small cell lung cancer. J Immunother Cancer. 2023 Aug;11(8):e006770. doi: 10.1136/jitc-2023-006770. PMID 37648263
- [Derived] Bratman SV, Yang SYC, Iafolla MAJ, Liu Z, Hansen AR, Bedard PL, Lheureux S, Spreafico A, Razak AA, Shchegrova S, Louie M, Billings P, Zimmermann B, Sethi H, Aleshin A, Torti D, Marsh K, Eagles J, Cirlan I, Hanna Y, Clouthier DL, Lien SC, Ohashi PS, Xu W, Siu LL, Pugh TJ. Personalized circulating tumor DNA analysis as a predictive biomarker in solid tumor patients treated with pembrolizumab. Nat Cancer. 2020 Sep;1(9):873-881. doi: 10.1038/s43018-020-0096-5. Epub 2020 Aug 3. PMID 35121950
- [Derived] Iafolla MAJ, Yang C, Chandran V, Pintilie M, Li Q, Bedard PL, Hansen A, Lheureux S, Spreafico A, Razak AA, Hakgor S, Giesler A, Pugh TJ, Siu LL. Predicting Toxicity and Response to Pembrolizumab Through Germline Genomic HLA Class 1 Analysis. JNCI Cancer Spectr. 2020 Dec 29;5(1):pkaa115. doi: 10.1093/jncics/pkaa115. eCollection 2021 Feb. PMID 33554038